CLINICAL TRIAL: NCT07256951
Title: Gen 2 Battrode Wear Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: BXU610410
Record Dates: First submitted 2025-11-21; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Adhesive Wear Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- adhesive one (Experimental)
  Interventions: Device: Adhesive
- Adhesive two (Experimental)
  Interventions: Device: Adhesive

INTERVENTIONS:
Device: Adhesive — 14 day wear

SUMMARY:
Validating adhesive wear time

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 18 years.
2. Completes the consent process as required.
3. Participants can speak and read English fluently.
4. Willing to allow shaving of device application area, as required.
5. Willing to take photos of the application area before wear, daily during wear, and immediately after removal.
6. Willingness to report current known pregnancy.

Exclusion Criteria:

1. Unable to comply with the study protocol and instructions for wearing the devices for up to 15 days.
2. Any pre-existing breached or compromised skin, skin rash, irritation or infection at the application area.
3. Any incision, wound or scar in the application area.
4. Participants with known skin allergies and sensitivities to adhesives.
5. Participants with scheduled electronic imaging (including magnetic resonance imaging), cardioversion, and/or procedures where device would be removed during the data collection period.
6. Participants with known history of cardiac arrhythmias.
7. Participants with chest anatomies not compatible with secure parasternal placement.
8. Use of clothing or garment that can dislodge or loosen the patch or bras with underwires or other worn items that might interfere with the devices under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Wear time | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Orange County Research Center, Lake Forest, California, United States